CLINICAL TRIAL: NCT02158117
Title: Bioavailability of a New Formulation of Nasal Naloxone for Prehospital Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPI-13-001
Record Dates: First submitted 2014-06-02; First posted 2014-06-06 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Drug Overdose
Keywords: Emergency Treatment; Morphine Derivates; Heroin; Antidotes; Administration, Intranasal
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nasal naloxone (Experimental): 8 and 16 mg/ml, comparator 1 mg/ml. Three daily occasions with at least 3 days washout between treatment (min 8 days).
  Interventions: Drug: nasal naloxone

INTERVENTIONS:
Drug: nasal naloxone — one puff in one nostril with the subject is lying down

SUMMARY:
Overdose with potential deadly outcome is a serious problem among opioid abusers, not least in Norway. The annual death toll from overdose is about 250, twice the annual death toll from traffic accidents. Those who inject heroin or other opioids are considered to have the highest risk for death from overdose. To save lives, immediate treatment with a μ-opioid antidote such as naloxone is required. Usually naloxone is injected into a muscle or a blood vessel. Administration of naloxone via the nose has been suggested as an alternative for use by emergency teams and possibly also bystanders. This is not only an easier way to give naloxone, but would also eliminate the risk for needle stick injuries and blood contamination. A pilot study in this hospital has shown no significant side effects or adverse reaction. While significant benefits are expected from developing an adequately formulated naloxone nasal spray for pre-hospital use, the risks to participants are minimal. Therefore this preclinical study in healthy volunteers will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal electrocardiogram (ECG)
* Hemoglobin: male 13.4 - 17.0 g/dL, female 11,7- 15.3 g/dL
* Creatinine: male 60- 105 micromol/L female 45- 90 micromol/L
* ASAT: male 15- 45 U/L, female 15- 35 U/L
* ALAT: male 10- 70 U/L female 10- 45 U/L
* Gamma GT: male 10- 80 U/L female 10- 45 U/L
* HCG normal under 3 ye/L
* Fertile women must use safe contraception and have a negative serum HCG at inclusion

Exclusion Criteria:

* Taking any medications including herbal medicines the last week prior to first treatment visit
* History of drug abuse
* History of prior drug allergy
* Having any local nasal disease or nasal surgery or recent cold for the last week
* Pregnancy
* Fertile women not using high efficacy contraceptives (Oral contraceptives, Patch (Evra), Implants, Vaginal ring, Hormonal IUD, Copper IUD, Sterilization) throughout the study period until their last visit.
* Lactating women
* Any reason why, in the opinion of the investigator, the patient should not participate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
bioavailability of naloxone | 2 weeks
  A LCMSMS method for determination of Naloxone in serum was developed using acetonitrile protein precipitation. Naloxone D5 was used as internal standard and quantitative determination was done by using Sciex Analyst version 1.5. The method is fully validated by assessing linearity, accuracy, precision, sensitivity, specificity/selectivity, in process and storage stability, dilution integrity and assay ruggedness according to Dadgar (1995) and Shah (1991). The method was found linear, accurate and precise across the dynamic range of 0.05 to 45 ng/ml. Limit of quantification (LOQ) was 0.05ng/ml with CV = 12.7% and inaccuracy < 7.8% (n = 17). Quality Controls (QC) in middle (n=18) and upper (n=18) calibration range had CV < 4.2% and inaccuracy <8.2 %

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) | 2 weeks
Time to maximum serum concentration (Tmax) | 2 weeks
adverse events | 2 weeks
  will be reported from the start of the first session to the follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Toril A Nagelhus Hernes, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

REFERENCES:
- [Result] Tylleskar I, Skulberg AK, Nilsen T, Skarra S, Jansook P, Dale O. Pharmacokinetics of a new, nasal formulation of naloxone. Eur J Clin Pharmacol. 2017 May;73(5):555-562. doi: 10.1007/s00228-016-2191-1. Epub 2017 Jan 31. PMID 28144724